CLINICAL TRIAL: NCT00002482
Title: A PHASE I-II TRIAL OF MUROMONAB (OKT-3) WITH LOW-DOSE CYCLOPHOSPHAMIDE
Brief Title: Monoclonal Antibody Plus Cyclophosphamide in Treating Patients With Metastatic Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Vincent Medical Center - Los Angeles (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000077247; SVMC-ONC-121; NCI-V90-0206
Record Dates: First submitted 1999-11-01; First posted 2004-06-28 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2007-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Immunization, Passive; Biological Therapy; Muromonab-CD3; Cyclophosphamide

INTERVENTIONS:
Biological: antibody therapy
Biological: biological therapy
Biological: muromonab-CD3
Drug: cyclophosphamide

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I/II trial to study the effectiveness of monoclonal antibody and cyclophosphamide in treating patients with metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the clinical feasibility and toxicity of monoclonal antibody OKT3 given with low-dose cyclophosphamide in patients with advanced malignancies. II. Perform serial immune monitoring on patients treated with this regimen. III. Identify any clinical responses produced by this regimen.

OUTLINE: Biological Response Modifier Therapy with Suppressor Cell Inhibition. Anti-CD3 Murine Monoclonal Antibody OKT3, MOAB OKT3; with Cyclophosphamide, CTX, NSC-26271.

PROJECTED ACCRUAL: At least 9 evaluable patients per diagnostic category will be required initially; if any response is seen during the dose-finding portion of the study, a total of 24 patients with that diagnosis will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Metastatic cancer considered incurable by standard therapy and for which no higher priority protocol is available Locally progressive primary brain tumors (e.g., astrocytoma, glioma) are also eligible Brain metastases allowed

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-4 (poor performance status brain tumor patients specifically eligible) Life expectancy: At least 2 months Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Pulmonary: No history of adult asthma No emphysema No pulmonary insufficiency No pulmonary edema Other: No AIDS or positive HIV serology No pregnant women

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1991-06

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Wiseman, MD, FACP, Study Chair
Locations (1):
- St. Vincent Medical Center - Los Angeles, Los Angeles, California, United States